CLINICAL TRIAL: NCT05113069
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of SHR-A1912 for Injection as Monotherapy in Patients With B-cell Lymphoma
Brief Title: A Study of SHR-A1912 for Injection in Patients With B Cell Lymphomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1912-I-101
Record Dates: First submitted 2021-11-05; First posted 2021-11-09 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: single arm for SHR-A1912
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): SHR-A1912
  Interventions: Drug: SHR-A1912

INTERVENTIONS:
Drug: SHR-A1912 — SHR-A1912, dose escalation and expansion.

SUMMARY:
To assess the safety and tolerability of SHR-A1912 in patients with B cell lymphoma, to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and recommended phase II dose (RP2D) of SHR-A1912.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to18 years old, male or female;
2. Eastern Cooperative Oncology Group (ECOG) performance status is 0 to 1;
3. Life expectancy >12 weeks;
4. Histologically or cytologically confirmed B cell lymphoma;
5. Relapsed and/or refractory disease after at least 1 prior treatment regimen;
6. At least one measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or one measurable extra nodal lesion, defined as > 1.0 cm in its longest diameter (no need for dose escalation stage).

Exclusion Criteria:

1. Received autologous stem cell transplantation within 12 weeks before the first study treatment; previously received allogeneic stem cell transplantation; received Car-T cell therapy within 12 weeks before the first study treatment;
2. History of recent major surgery or severe trauma within 4 weeks before the first study treatment;
3. Received anti-tumour treatment within 2 weeks before the first study treatment;
4. Central nervous system (CNS) infiltration;
5. Active infection with HBV or HCV;
6. History of immunodeficiency, including HIV serotest positive, or other acquired or congenital immunodeficiency diseases, and active tuberculosis;
7. Active infection or unexplained fever>38.5℃;
8. History of severe cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 21 Days after the 1st dosing (first cycle)
Dose Limited Toxicity (DLT) | 21 Days (first cycle)
Maximum tolerable dose (MTD) | 21 Days (first cycle)
Recommended phase II dose (RP2D) | Up to approximately 2 years

SECONDARY OUTCOMES:
Adverse Events | 12 weeks after the last dose
Time of maximum observed plasma concentration (Tmax) of SHR-1912 | 21 days after last dose
Maximum observed plasma concentration (Cmax) of SHR-1912 | 21 days after last dose
Area under the plasma concentration time curve (AUC) of SHR-1912 | 21 days after last dose
Anti-drug antibody (ADA) of SHR-A1912 | 12 weeks after last dose
Complete Response Rate (CR) | Up to approximately 2 years
Objective Response Rate (ORR) | Up to approximately 2 years
Duration of Response (DoR) | Up to approximately 2 years
Disease Control Rate (DCR) | Up to approximately 2 years
Progression-Free Survival (PFS) | Up to approximately 2 years
Overall Survival (OS) | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided